CLINICAL TRIAL: NCT02203292
Title: Transfusion Requirements After Head Trauma
Acronym: TRAHT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, André Luiz Nunes Gobatto, M.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32520914.3.0000.0068
Record Dates: First submitted 2014-07-27; First posted 2014-07-29 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Blood Transfusion
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal (Active Comparator): Liberal transfusion strategy. Patients will have red blood cells transfused only if Hb < 9.0 g/dL
  Interventions: Behavioral: Liberal transfusion strategy
- Restrictive (Experimental): Restrictive transfusion strategy. Patients will have red blood cells transfused only if Hb < 7.0 g/dL
  Interventions: Behavioral: Restrictive transfusion strategy

INTERVENTIONS:
Behavioral: Liberal transfusion strategy — Patients will have red blood cells transfused only if Hb < 9.0 g/dL
  Arms: Liberal
Behavioral: Restrictive transfusion strategy — Patients will have red blood cells transfused only if Hb < 7.0 g/dL
  Arms: Restrictive

SUMMARY:
TRAHT is a pilot randomized clinical trial designed to evaluate safety and feasibility of two red blood cells transfusion thresholds in moderate or severe traumatic brain injured patients

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Moderate or severe traumatic brain injury, defined as Glasgow coma scale less than or equal to 12 at hospital admission
* Hemoglobin lower than 9.0 g/dL within 7 days from hospital admission

Exclusion Criteria:

* Glasgow coma scale equal to 3 with dilated pupils bilaterally
* Previous neurological sequelae
* Pregnant women
* Jehovah's Witnesses
* Hemorrhagic shock at randomization
* Moribund patients
* Unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin difference | 14 days
  Hemoglobin difference between restrictive and liberal groups

SECONDARY OUTCOMES:
Number of transfused patients | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Number of red blood cell packages transfused | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
ICU mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Hospital mortality | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
180 days mortality | Participants will be followed for 180 after hospital discharge
Blood stream infection | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Positive blood culture with a pathogenic microorganism
Re-bleeding | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Intensity of measures to reduce intracranial pressure | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Measures to reduce intracranial pressure such as sedation, hypertonic solutions, hypothermia, liquorice drainage, decompressive craniectomy or hyperventilation
Hospital length of stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
ICU length of stay | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Mechanical ventilation free days | 28 days
  Days breathing without assistance from hospital admission to day 28.
Extended Glasgow Outcome Scale at hospital discharge | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Extended Glasgow Outcome Scale after 6 months | 180 days
Myocardial Infarction | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Acute Respiratory Distress Syndrome | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Septic Shock | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
Cerebral autoregulation | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Cerebral autoregulation as measure by the transcranial doppler
Pulsatility index | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Pulsatility index as measure by the transcranial doppler

CONTACTS AND LOCATIONS:
Overall Officials: André LN Gobatto, M.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Gobatto ALN, Solla D, Brasil S, Taccone FS, Carlotti CG Jr, Malbouisson LMS, Paiva WS. Progressive hemorrhagic injury and ischemia after severe traumatic brain injury according to hemoglobin transfusion thresholds: a post-hoc analysis of the transfusion requirements after head trauma trial. Crit Care. 2024 Jul 3;28(1):218. doi: 10.1186/s13054-024-04981-5. No abstract available. PMID 38961443
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Gobatto ALN, Link MA, Solla DJ, Bassi E, Tierno PF, Paiva W, Taccone FS, Malbouisson LM. Transfusion requirements after head trauma: a randomized feasibility controlled trial. Crit Care. 2019 Mar 12;23(1):89. doi: 10.1186/s13054-018-2273-9. PMID 30871608